CLINICAL TRIAL: NCT01150864
Title: Effects of Airway Conditioning Devices on Ventilator Associated Pneumonia:a Randomized Clinical Trial
Acronym: AirconVAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Paolo Severgnini, MD, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0001069
Record Dates: First submitted 2010-05-24; First posted 2010-06-25 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Acute Lung Injury
Keywords: Hot water humidifier, Passive heat and moisture exchangers
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Passive Humidifier (Active Comparator): The Passive Humidifier (HME)will changed every 24 hours
  Interventions: Device: Airway Conditioning
- Active-Passive humidifier (Active Comparator): The Active-Passive Humidifier will be changed every 24 hours
  Interventions: Device: Airway Conditioning
- Hot Water Humidifier (Active Comparator): Hot water humidifier will be set at 36-37 °C
  Interventions: Device: Airway Conditioning

INTERVENTIONS:
Device: Airway Conditioning — Each Passive device will be changed daily. When using Active and Passive devices as well as Active-Passive devices the ventilatory circuit will be changed every 7 days.
  Other Names: Passive: Hygrobac; Active-Passive: Hygrovent Gold; Hot Water: Tyco HC 2000 heated wire

SUMMARY:
The main hypothesis are:

1. Passive and Active-Passive airway conditioning devices reduce the incidence of ventilator associated pneumonia
2. Active-Passive airway conditioning devices reduce the incidence of endotracheal tube obstruction
3. Nurses' workload is reduced with Passive and Active-Passive airway conditioning devices

DETAILED DESCRIPTION:
For all Three lines of the study we record Clinical Pulmonary Infection score and Airways Care Score, SOFA (Sequential Organ Failure Assessment), sedation strategy, Glasgow Coma Score and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients mechanically ventilated with PaO2/FiO2 lower than 300
* Age higher than 18 years
* Invasive mechanical ventilation
* Endotracheal intubation or tracheostomy for more than 24 hours

Exclusion Criteria:

* Non invasive ventilation
* Severe ARDS (PaO2/FiO2 lower than 100, or PaCO2 higher than 60 mmHg)
* Inefficient cough
* Head Trauma
* Spinal cervical trauma
* Chest trauma
* Pregnancy
* Expectance of poor survival within 72 hours
* Congenital airway disease
* Immunosuppression
* Supraglottic aspiration devices

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2010-04; Primary Completion 2015-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Reduction of ventilator associated pneumonia | 2 years
  development of ventilator associated pneumonia after 48 hours of mechanical ventilation

SECONDARY OUTCOMES:
Endotracheal tube obstruction | 2 years
  difficulties to introduce the airway suction catheter and or need to change the tracheal tube
nurses' workload | 2 years
  time spent at the bedside by nurses to clear airway's secretions and or to remove water condense from ventilatory circuit

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pelosi, MD, Study Director — Universita' degli Studi dell'Insubria, Varese, Italy; Paolo Severgnini, MD, Principal Investigator — University of Insubria, Varese, Italy
Locations (1):
- Ospedale di Circolo, Varese, Italy